CLINICAL TRIAL: NCT03390387
Title: Moscow-Berlin 2015 Multicenter Randomized Study for Treatment of Acute Lymphoblastic Leukemia in Children, Adolescents and Young Adults
Brief Title: Childhood Acute Lymphoblastic Leukemia Treatment Protocol Moscow-Berlin 2015 (ALL-MB 2015)
Acronym: ALL-MB 2015
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Principal Investigator, Karachunskiy Alexander, Deputy director - Director of Institute of Oncology, Radiology and Nuclear Medicine of Federal Research Institute of Pediatric hematology, Oncology and Immunology, Federal Research Institute of Pediatric Hematology, Oncology and Immunology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALL-MB 2015
Record Dates: First submitted 2017-12-27; First posted 2018-01-04 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Childhood Acute Lymphoblastic Leukemia
Keywords: Acute lymphoblastic leukemia, children, adolescents, treatment
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Dexamethasone; Methylprednisolone; Daunorubicin; Idarubicin; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Dexa intermittent (Experimental): Induction therapy with intermittent Dexamethasone administration (1-15 days - 6 mg/m2, 15-22 day - pause, 22-29 days - 6 mg/m2).
  Interventions: Drug: Dexamethasone intermittent
- Dexa constant (Active Comparator): Induction therapy with continuous Dexamethasone administration (6 mg/m2 1-29 days).
  Interventions: Drug: Dexamethasone continuous
- Dexa (Active Comparator): Therapy with Dexamethasone (6 mg/m2) as basic glucocorticoid preparation.
  Interventions: Drug: Dexamethasone
- Medrol (Experimental): Therapy with Methylprednisolone (60 mg/m2) as basic glucocorticoid preparation.
  Interventions: Drug: Methylprednisolone
- IDA (Experimental): Induction and consolidation therapy with Idarubicin
  Interventions: Drug: Idarubicin
- DNR (Active Comparator): Induction and consolidation therapy with Daunorubicin
  Interventions: Drug: Daunorubicin
- Protocol Ib+ (Experimental): Two-phase induction therapy (additional second phase of induction - protocol Ib)
  Interventions: Drug: Second phase of induction
- Protocol Ib- (Active Comparator): Standard induction therapy (without second phase)
  Interventions: Drug: Standard induction therapy
- Bortezomib- (Active Comparator): Consolidation therapy without Bortezomib
  Interventions: Drug: Standard consolidation therapy
- Bortezomib+ (Experimental): Consolidation therapy with Bortezomib 1.3 mg/m2 N12 (N4 in each reinduction)
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Dexamethasone continuous — 6 mg/m2, per os, in two divided doses per day q12 hours. 1-28 day (dose in the first few days is depending on the total tumor mass). From day 29 the dose of dexamethasone is reducing: days 29-31 - 3 mg/m2, days 32-34 - 1.5 mg/m2, days 35-36 - 0.75 mg/m2; then dexamethasone is discontinued completely.
  Arms: Dexa constant
Drug: Dexamethasone intermittent — 6 mg/m2, per os, in two divided doses per day q12 hours. Days: 1-14 (dose in the first few days is depending on the total tumor mass) and 22-28; days 15-21 - pause. From day 29 the dose of dexamethasone is reducing: days 29-30 - 3 mg/m2, days 31-32 - 1.5 mg/m2, then dexamethasone is discontinued completely.
  Arms: Dexa intermittent
Drug: Dexamethasone — Induction: 6 mg/m2, per os, in two divided doses per day q12 hours. 1-28 day (dose in the first few days is depending on the total tumor mass). From day 29 the dose of dexamethasone is reducing: days 29-31 - 3 mg/m2, days 32-34 - 1.5 mg/m2, days 35-36 - 0.75 mg/m2; then dexamethasone is discontinued completely.
  Consolidation: 6 mg/m2 per os, in two divided doses per day q12 hours. Weeks 13-14 (days 85-98), weeks 21-22 (days 141-154), weeks 29-30 (days 197-210), weeks 37-38 (days 253-260), weeks 45-46 (days 309-316), weeks 53-54 (days 365-372).
  Maintenance therapy: 6 mg/m2, per os, in two divided doses per day q12 hours, for 10 days followed by quick discontinuation during 3 days. Weeks 61-62, 69-70, 77-78, 85-86, 93-94.
  Arms: Dexa
Drug: Methylprednisolone — Induction: 60 mg/m2, per os, in two divided doses per day q12 hours. 1-28 day (dose in the first few days is depending on the total tumor mass). From day 29 the dose of dexamethasone is reducing: days 29-31 - 30 mg/m2, days 32-34 - 15 mg/m2, days 35-36 - 8 mg/m2; then methylprednisolone is discontinued completely.
  Consolidation: 60 mg/m2 per os, in two divided doses per day q12 hours. Weeks 13-14 (days 85-98), weeks 21-22 (days 141-154), weeks 29-30 (days 197-210), weeks 37-38 (days 253-260), weeks 45-46 (days 309-316), weeks 53-54 (days 365-372).
  Maintenance therapy: 60 mg/m2, per os, in two divided doses per day q12 hours, for 10 days followed by quick discontinuation during 3 days. Weeks 61-62, 69-70, 77-78, 85-86, 93-94.
  Arms: Medrol
Drug: Daunorubicin — Induction: 45 mg/m2, intravenously, for 6 hours on days 8 and 22. Consolidation: 30 mg/m2, intravenously, for 6 hours on days 44, 65 (consolidation S1); 107, 121 (consolidation S2); and 163 (consolidation S3).
  Arms: DNR
Drug: Idarubicin — Induction: 10 mg/m2, intravenously, for 6 hours on days 8 and 22. Consolidation: 8 mg/m2, intravenously, for 6 hours on days 44, 65 (consolidation S1); 107, 121 (consolidation S2); and 163 (consolidation S3).
  Arms: IDA
Drug: Bortezomib — 1.3 mg/м2, intravenously, bolus injection. Days 85, 89, 92, 96 (consolidation S1); 141, 145, 148, 152 (consolidation S2) and 197, 201, 204, 208 (consolidation S3).
  Arms: Bortezomib+
Drug: Second phase of induction — Cyclophosphamide (1,000 mg/m2, intravenously, for 1 hour - days 43 and 71); Cytarabine (75 mg/m2/day, intravenously, bolus injection. Four blocks of 4 days each, days 46-48, 52-55, 59-62, and 66-69); 6-mercaptopurine (60 mg/m2/day, per os, days 43-71); Triple intrathecal therapy (days 52 and 66)
  Arms: Protocol Ib+
Drug: Standard induction therapy — Dexamethasone (6 mg/m2, p/o; 1-29 days); Daunorubicin (45 mg/m2, i.v.; day 8 and 22); Vincristine (1.5 mg/m2, i.v.; days 8, 15, 22, 29 and 36); Triple intrathecal therapy (Methotrexate/Cytarabine/Prednisone; days 0/1, 8, 15, 22, 29 and 36)
  Arms: Protocol Ib-
Drug: Standard consolidation therapy — Consolidation consists of 3 phases: S1, S2 and S3. Each phase is a 6-week therapy with 6-mercaptopurine (50 mg/m2 per day, daily, orally), methotrexate (30 мг/м2, i.m., weekly) and L-asparaginase (10 000 U/m2, i.m., weekly), followed by 2 weeks of re-induction with Vincristine (1.5 mg/m2, i.v., days 1 and 8 of reinduction) plus Dexamethasone (6 mg/m2, p/o, daily, for 10 days followed by quick discontinuation during 3 days). Daunorubicin (30 mg/м2, i.v., N2 during S1, N2 during S2 and N1 during S3). Triple intrathecal therapy (Methotrexate/Cytarabine/Prednisone) N12 (4 injections per each phase)
  Arms: Bortezomib-

SUMMARY:
QUESTIONS AND OBJECTIVES OF ALL-MB 2015 STUDY

1. Will the new risk group stratification (especially of T-ALL) to improve overall and event-free survival?
2. Will the new protocol is effective and feasible in patients older than 15 years, and especially in young adults?
3. Whether the intermittent dexamethasone administration in induction will result in a decrease in toxicity and mortality without loss of efficacy?
4. Whether the methylprednisolone administration as basic glucocorticoids during induction, consolidation and maintenance therapy will lead to decrease of severe infections and early mortality rate, improve survival and therapy compliance in adolescents and young adults with B-precursor ALL?
5. Whether the administration of Bortezomib in patients with B-precursor ALL with initial WBC≥100,000/µl will improve treatment outcome?
6. Whether the administration of Idarubicin instead Daunorubicin in low-risk T-ALL patients and two-phase induction in intermediate-risk T-ALL patients will reduce relapse rate and improve survival?

ELIGIBILITY:
Inclusion Criteria:

* Age at diagnosis at 1 to 50 years.
* The start of induction therapy within a time interval of study recruitment phase.
* The diagnosis of ALL is to be proved by the morphological, cytochemical, and immunological analysis of tumor cells in bone marrow (see "Diagnostics"). Patients with B-cell (Burkitt) ALL are excluded.
* Informed consent of the patient parents (guardians) to be treated in one of the clinics included in this multicenter study.

Exclusion Criteria:

* ALL is a second malignancies;
* The disease is a relapse of previously misdiagnosed and, therefore, inadequately treated ALL;
* There is severe concomitant disease, which significantly impedes chemotherapy protocol (such as multiple malformations, heart diseases, metabolic disorders, etc.);
* There is a lack of important data needed for the exact adherence to the cytostatic therapy according to a specific chemotherapy protocol (differential diagnosis of ALL-AML (acute myeloid leukemia) is not possible, stratification according to therapeutic group is not possible);
* The patient was treated before for a long time with cytotoxic drugs;
* There were treatment deviations not covered by the protocol and/or not due to side effects of treatment and/or complications of the disease

Ages: 1 Year to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4000 (Estimated)
Dates: Start 2015-11 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | 3 years, 5 years and 10 years after study start
Overall survival | 3 years, 5 years and 10 years after study start
Cumulative incidence of relapse | 3 years, 5 years and 10 years after study start

SECONDARY OUTCOMES:
Early death rate | 3 years, 5 years and 10 years after study start
Remission death rate | 3 years, 5 years and 10 years after study start

CONTACTS AND LOCATIONS:
Overall Officials: Alexander I. Karachunskiy, Professor, MD, Principal Investigator — Research Institute of Pediatric Hematology, Oncology and Immunology
Locations (58):
- prof. R.O.Eolyan Hematology Center, Yerevan, Armenia
- Belarus (3):
  - Republican Research and Practical Center of Radiation Medicine and Human Ecology, Homyel
  - Republic Research and Practical Center of Pediatric Oncology, Hematology and Immunology, Minsk
  - Mogilev Regional Children's Hospital, Mogilev
- National Oncology and Hematology Center, Ministry of Health of the Kyrgyz Republic, Bishkek, Kyrgyzstan
- Russia (52):
  - Arkhangelsk Regional Clinical Children's Hospital, Arkhangelsk
  - Regional Clinical Children's Hospital, Astrakhan
  - Altay Regional Clinical Children's Hospital, Barnaul
  - Amur Regional Clinical Children's Hospital, Blagoveshchensk
  - Bryansk Regional Children's Hospital, Bryansk
  - Chelyabinsk Regional Clinical Children's Hospital, Chelyabinsk
  - Transbaikal Regional Oncology Dispensary, Chita
  - Irkutsk Regional Children Clinical Hospital, Irkutsk
  - Ivanovo Regional Clinical Hospital, Ivanovo
  - Republic Clinical Children's Hospital, Izhevsk
  - Regional Clinical Children's Hospital, Khabarovsk
  - Kirov Research Institute of Hematology and Blood Transfusion, Kirov
  - Regional Clinical Children's Hospital, Krasnodar
  - Krasnoyarsk Territorial Clinical Children's Hospital, Krasnoyarsk
  - Kurgan Regional Clinical Children's Hospital, Kurgan
  - Regional Clinical Children's Hospital, Kursk
  - Regional Children's Hospital, Lipetsk
  - Republic Children's Clinical Hospital, Makhachkala
  - Morozov Children's Municipal Clinical Hospital, Moscow
  - Research Institute of Pediatric Hematology, Oncology and Immunology named after Dmitry Rogachev, Moscow
  - Russian Children's Clinical Hospital, Moscow
  - Murmansk Clinical Children's Hospital, Murmansk
  - Republic Clinical Children's Hospital, Nal'chik
  - Nizhnevartovsk Regional Clinical Children's Hospital, Nizhnevartovsk
  - Regional Clinical Children's Hospital, Nizhny Novgorod
  - Novokuznetsk Municipal Clinical Children's Hospital N4, Novokuznetsk
  - Novosibirsk Central District Clinical Hospital, Novosibirsk
  - Orenburg Regional Clinical Oncology Dispensary, Orenburg
  - Regional Clinical Children's Hospital, Oryol
  - Perm Territorial Clinical Children's Hospital, Perm
  - Regional Clinical Children's Hospital, Rostov-on-Don
  - Rostov Research Institute of Oncology, Rostov-on-Don
  - N. Dmitrieva Ryazan Regional Clinical Children's Hospital, Ryazan
  - Almazov National Medical Research Center, Saint Petersburg
  - Children's Municipal Hospital N1, Saint Petersburg
  - Municipal Clinical Hospital N31, Saint Petersburg
  - N.N.Petrov National Medical Research Oncology Center, Saint Petersburg
  - R. Gorbacheva Research Institute of Pediatric Hematology and Transfusiology; Pavlov First Saint-Petersburg State Medical University, Saint Petersburg
  - Municipal Clinical Children's Hospital N1, Samara
  - Regional Children's Clinical Hospital, Stavropol
  - Surgut Regional Clinical Hospital, Surgut
  - Republic Clinical Children's Hospital, Syktyvkar
  - Tomsk Regional Clinical Hospital, Tomsk
  - Tula Regional Clinical Children's Hospital, Tula
  - Republic Clinical Children's Hospital, Ulan-Ude
  - Ulyanovsk Regional Children's Clinical Hospital, Ulyanovsk
  - Regional Children's Clinical Hospital N1, Territorial Children's Hematological Center, Vladivostok
  - Vologda Regional Clinical Children's Hospital, Vologda
  - Voronezh Regional Clinical Children's Hospital N1, Voronezh
  - Republic Hospital N1 - National Medicine Centre, Yakutsk
  - Regional Clinical Children's Hospital, Yaroslavl
  - Regional Clinical Children's Hospital N1; Children Oncology and hematology Center, Yekaterinburg
- Research Institute of Hematology and Blood Transfusion, Tashkent, Uzbekistan

REFERENCES:
- See also: Study web-site — http://www.mbstudy.net